CLINICAL TRIAL: NCT07183527
Title: Hybrid Type I Effectiveness-Implementation Cluster Randomized Trial of CARES
Brief Title: Hybrid Type I Effectiveness-implementation Cluster Randomized Controlled Trial of CARES
Acronym: CARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Steel, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY24070065; 1R01CA296402 (NIH)
Record Dates: First submitted 2025-08-22; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: CARES; Standard of Care
Keywords: implementation; stepped collaborative care; integrated screening and treatment; cluster randomized controlled trial; cancer; screening
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARES (Experimental): Integrated Screening and Stepped Collaborative Care Intervention
  Interventions: Behavioral: CARES
- Standard of Care (SOC) (Active Comparator): Integrated screening and referred to treatment in the community and/or at the cancer center
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: CARES — Integrated screening and stepped collaborative care
  Arms: CARES
Behavioral: Standard of Care (SOC) — Screening and referral of patient to provider in the community or cancer center
  Arms: Standard of Care (SOC)

SUMMARY:
The trial will examine the effectiveness and facilitators and barriers of implementation of CARES, an integrated screening and stepped collaborative care intervention

DETAILED DESCRIPTION:
Over 18 million Americans are living with cancer. Half of them report clinically significant levels of depression, pain, and/or fatigue. According to the NIH consensus statement, these are the three most common and distressing cancer-related symptoms. These symptoms lead to poorer health-related quality of life (HRQoL) and cancer-related treatment adherence, higher unplanned health care utilization and costs, and reduced life expectancy.

Investigators observed in a trial of CARES, an integrated screening and stepped collaborative care intervention, that 75% versus 4% of participants initiated treatment when compared to standard of care. Improvements in HRQoL and reductions in pain, depression, fatigue, emergency room visits, readmissions to the hospital, and length of stay in the hospital were observed. The cost savings to the health care system was $17,085 per patient per year when compared to standard of care.

The overarching objective of the proposed study is to move CARES from research to routine clinical care. Investigators plans to test the effectiveness of CARES in a pragmatic trial or "real world" setting. An implementation-focused process evaluation of participant and clinician engagement with CARES guided by the RE-AIM framework will also be performed. Finally, to prepare to disseminate the intervention, a full cost-effectiveness analysis of CARES will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cancer
* Age 18 years or older
* Read and write in English

Exclusion Criteria:

* Evidence of thought disorder
* Evidence of delusions
* Evidence of hallucinations
* Evidence of suicidal ideation with a plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2030-01-10 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-General | Enrollment to the end of study for participant (12 months). The primary time point is 6 months
  Health Related Quality of Life. A total score (0-108) and subscales scores (0-24 or 0-28) with a higher score reflecting a better quality of life
Functional Assessment of Cancer Therapy-General | Enrollment to the end of study for participant (12 months). The 12 months outcome will be a measure of maintenance of benefits.
  Health Related Quality of Life. A total score (0-108) and subscales scores (0-24 or 0-28) with a higher score reflecting a better quality of life

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Screening to baseline and baseline to 12 months. The primary outcome will be at 6-months.
  Depressive Symptoms. A higher score reflecting more severe depressive symptoms (range of scores 0-27)
Brief Pain Inventory. | Screening to baseline and baseline to 12 months. The primary outcome will be from baseline to 6-months
  Pain intensity and interference. The Pain, Enjoyment, and General Activity score (0-10) will be used as the secondary outcome. A higher score reflects greater pain interference.
Generalized Anxiety Disorder -7 | Screening to baseline and baseline to 12 months. The primary time point is from baseline to 6 months.
  Anxiety. The total score ranges from 0-21. A higher score indicates higher levels of anxiety.
FACIT Fatigue | Baseline to 12 months. The primary time point will be 6 months.
  Fatigue. A total score ranges from 0-52. A higher score indicates less fatigue.
PROMIS Depression | Baseline to 12 months. The primary time point is 6 months. The questionnaire will be used for treatment response 0-24 weeks (every 4 weeks).
  Depressive symptoms. The range is from a T scores of 0-100 with a higher score reflecting higher levels of depressive symptoms.
PROMIS Anxiety | Baseline to 12 months.
  Anxiety. Scores range from a T score of 0-100 and a higher score reflects worse anxiety. Used for treatment response and primary endpoint 6 months.
Fatigue Assessment Scale | Enrollment to the end of study for participant (12 months). The primary time point is 6 months. The questionnaire will also be used for treatment response 0-24 weeks (every 4 weeks).
  Fatigue. The total score ranges from 10 to 50. A higher score reflects more severe fatigue.
Pain Visual Analog Scale | Baseline to 12 months. The 6 month time point is primary. The questionnaire will also be used for treatment response 0-24 weeks (every 4 weeks) and then for the booster session at the end of treatment up until 12 months.
  Pain Severity. Total score ranges from 0-100. A higher score reflects higher levels of pain.
Pittsburgh Sleep Quality Index | Enrollment to the end of study for participant (12 months). The primary time point is 6-months.
  Sleep problems. The total sleep quality (0-21) and subscales including the sleep duration (0-24), sleep disturbance (0-3), sleep latency (0-3), days of dysfunction (0-3), efficiency (0-3), overall sleep quality (0-3), medications to sleep (0-3). A higher score means more sleep problems.
Interpersonal Support Evaluation List | Enrollment to the end of study for participant (12 months). The primary time point is 6-months.
  Social support. A higher score reflects better social support. The range of scores 0-48 with subscales including appraisal (0-16), belonging (0-16), and tangible (0-16).
Patient Health Questionnaire-9 | Screening to baseline and baseline to 12 months. The 12 months outcome will be a measure of maintenance of benefits.
  Depressive Symptoms. Scores range from 0-27 with a higher score reflecting higher levels of depressive symptoms
Brief Pain Inventory. | Screening to baseline and baseline to 12 months. The 12 month PEG score will reflect maintenance of treatment.
  Pain intensity and interference. The Pain, Enjoyment, and General Activity score (0-10) will be used as the secondary outcome. A higher score reflects greater pain interference.
Generalized Anxiety Disorder -7 | Screening to baseline and baseline to 12 months. The 12 months time point will assess maintenance of change.
  Anxiety. The total score ranges from 0-21. A higher score indicates higher levels of anxiety.
FACIT Fatigue | Enrollment to the end of study for participant (12 months). The 12 months time point will reflect maintenance of change in fatigue.
  Fatigue. A total score ranges from 0-52. A higher score indicates less fatigue.
COST | Enrollment to the end of study for participant (12 months). The primary time point will be at 12 months.
  Financial toxicity. The range of scores is from 0-44 and a higher scores reflects a better financial well being.
Cost Coping | Enrollment to the end of study for participant (12 months). The primary time point will be 12 months.
  Cost coping strategies. The total score is the number of cost coping strategies a patient uses to manage their financial costs associated with their medical care. The total number of cost coping strategies is 0-26.
EQ 5D 5L (this is the title of the instrument there is no non abbreviated title) | Enrollment to the end of study for participant (12 months). The primary time point is 12 months.
  Health related quality of life. Total score ranges from 0-25 for part 1 and 0 to 100 for part 2. A higher score reflects a better quality of life.
Cost Assessment | Enrollment to the end of study for participant (12 months). The primary time point is 12 months.
  Health Care Utilization. There is no total score for this questionnaire as it will be used to estimate costs.
PROMIS Depression | Enrollment to the end of study for participant (12 months). The 12 month time point will be used to assess maintenance of change.
  Depressive symptoms. The range is from 0-100 with a higher score reflecting higher levels of depressive symptoms.
PROMIS Anxiety | Enrollment to the end of study for participant (12 months). The 12 months time point is to assess maintenace of change.
  Anxiety. Scores range from 0-100 and a higher score reflects worse anxiety.
Fatigue Assessment Scale | Enrollment to the end of study for participant (12 months). The 12 months time point will assess maintenance of change.
  Fatigue. The total score ranges from 10 to 50. A higher score reflects more severe fatigue.
Pain Visual Analog Scale | Enrollment to the end of study for participant (12 months). The 12 months time point is to assess maintenance of change.
  Pain Severity. Total score ranges from 0-100. A higher score reflects higher levels of pain.
Pittsburgh Sleep Quality Index | Enrollment to the end of study for participant (12 months). The 12 months time point is to assess maintenance of change.
  Sleep problems. The total sleep quality (0-21) and subscales including the sleep duration (0-24), sleep disturbance (0-3), sleep latency (0-3), days of dysfunction (0-3), efficiency (0-3), overall sleep quality (0-3), medications to sleep (0-3). A higher score means more sleep problems.
Interpersonal Support Evaluation List | Enrollment to the end of study for participant (12 months). The 12-month time point will assess maintenance of change
  Social support. A higher score reflects better social support. The range of scores 0-48 with subscales including appraisal (0-16), belonging (0-16), and tangible (0-16).
Activity Based Costs | Enrollment to the end of study for participant (12 months). The primary time point is 12 months.
  Health care costs. Range could be 0 to 10 million dollars
Adherence to outpatient appointment | Enrollment to the end of study for participant (12 months). The primary time point is 12 months.
  Adherence to outpatient appointments. Percent of appointments missed out of total appointment in 12 months.
Complications | Baseline to 12 months
  Number of complications from procedures or surgeries during 12 months post randomization. The primary time point is 12 months.
Length of Stay in the Hospital | Baseline to 12 months
  Number of days patient was in the hospital. The primary end point is 12 months
Emergency Room Visits | 12 months
  Number of emergency room visits in 12 months post-randomization. The primary end point is 12 months
30-day readmissions | Baseline to 12 months
  Unplanned readmission to the hospital after a procedure or surgery within 30 days. Primary end point 12 months
90-day readmission | Baseline to 12 months
  Unplanned readmission to the hospital after a procedure or surgery within 90 days. The primary endpoint is 12 months
PROMIS Fatigue | Screening to baseline and baseline to 12 months
  Assesses fatigue in cancer patients. Higher score reflects greater fatigue. Score range from a T score 0-100. Primary end point baseline to 6 months
PROMIS Fatigue | Screening to baseline and baseline to 12 months
  Assesses fatigue in cancer patients. Higher score reflects greater fatigue. Score range from a T score 0-100. Secondary endpoint 12 months

OTHER OUTCOMES:
Modified Adverse Childhood Events | The questionnaire will only be administered at baseline
  Adverse events in childhood. The total score ranges from 0-16. A higher score reflects a greater number of early adverse events.
Sociodemographic factors | Administered at baseline only.
  Sociodemographic characteristics of patient (e.g., age, sex, race, ethnicity, etc). No total score.
Adherence to experimental treatment | Baseline to 12 months
  Patient adherence to intervention. Reported as percent completed out of prescribed number of sessions (6-24).
Adherence to Boosters | Baseline to 12 months
  Number of booster sessions completed.
Adherence to home practice | Enrollment to end of study (12 months).
  Patient adherence to intervention. Reported as percent completed.
Height | Baseline through 12 months
  Height in inches
Weight | Baseline to 12 months
  Weight in pounds
Body Mass Index | Baseline to 12 months
  703 x weight x height x 2
Psychiatric diagnoses | Baseline to 12 months
  The measure will provide information that is self-reported by the patient about any new diagnoses (e.g., depression, anxiety). No total score. Frequency of psychiatric diagnoses
Psychiatric or Psychological Treatments | Baseline to 12 months
  The treatments the person may have sought (e.g., counseling, medication, support group, pain clinic, palliative care). No total score. Frequency of treatments patients sought for symptoms
Patient cancer diagnosis | Baseline to 12 months
  Patient cancer diagnoses
Cancer treatments | Prior treatments before baseline and baseline to 12 months
  Past cancer treatments (e.g., surgery, chemotherapy, immunotherapy). No total score. Frequency of treatments.
Stage of Cancer | at diagnosis and changes from baseline to 12 months
  Stage of cancer
Routine laboratory values | Baseline 12 months
  Routine laboratory values (e.g., CEA, WBC, RBC)
Medical comorbities | Prior to baseline and baseline to 12 months
  Medical comorbidities (e.g., hypertension, diabetes). Total number and Charlson Comorbidly Index
Medications | Prior to baseline and baseline to 12 months
  Medications (e.g., antihypertensives, antidepressants). Number of medications, dose of medication, type of medication, and prescriber
Disease progression | Baseline to 12 months
  Disease progression. Measured by Complete response, partial response, disease progression, or stable disease
Residential Segregation | Baseline to 12 months
  Segregation as measured by publicly available resources and mapped based on the United States Census geographic identifiers
Gini Index | Baseline to 12 months
  Income inequality measured using publicly available resources and mapped based on the United States Census geographic identifiers
National Walkability | Baseline to 12 months
  Walkability of neighborhood based on publicly available resources and mapped based on the United States Census geographic identifiers
Area Deprivation Index | Baseline to 12 months
  Socioeconomic disadvantage as measured by publicly available resources and mapped based on the United States Census geographic identifiers
Rural Urban Continuum Code | Baseline to 12 months
  Measure of the rural versus urban residence. Measured using publicly available resources and mapped based on the United States Census geographic identifiers
Intervention Delivery | Baseline to 12 months
  How the intervention was delivered (e.g., phone, videoconference, face to face)
Patient location at time of intervention | Baseline to 12 months
  Where the patient was located when receiving the intervention
Session Content | Baseline to 12 months
  What session content the patient received (e.g., monitoring automatic thoughts, sleep hygiene, energy conservation strategies).
Homework completion | Baseline to 12 months
  Where and what homework was completed. Number of homework assignments and location of completion (e.g., home or in session)
Patient engagement with intervention content | Baseline to 12 months
  Therapists' ratings of patient engagement with the session material. 7 point Likert scale
Patient engagement with homework | Baseline to 12 months
  Therapist reported patient engagement with homework. Likert scale 1-7
Patient-Therapist Rapport | Baseline to 12 months
  Therapist rating of patient-therapist rapport. 1-7 Likert Scale
Crisis intervention | Screening to 12 months
  Number of patients reporting suicidal ideation and plan during screening and treatment. Number of patients requiring crisis intervention.
Change in Medication for Symptoms | Baseline to 12 months
  Initiation or change in medication dose, frequency, type, and health care provider who changed or initiated medication as reported by the patient and verified by medical record.
Symptoms at Screening | Screening to 12 months
  The number of patients who screened negative and positive for anxiety, depressive symptoms, fatigue, and pain

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Steel, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center (UPMC) Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be placed in data repository
Time Frame: After final outcomes are reported in published format
Access Criteria: Qualified researchers with aims and hypotheses that are approved by the study team